CLINICAL TRIAL: NCT03478254
Title: Adherence to Guidelines for Influenza, Pneumococcal and Hepatitis B Vaccination in Adult Patients With Type 1 Diabetes Mellitus (AVADI-1).
Brief Title: Adherence to Guidelines VAccination in Type 1 DIabetes Mellitus Patients (AVADI-1).
Acronym: AVADI-1
Status: Completed | Type: Observational
Sponsor: Jesús Moreno Fernández (Other)
Collaborators: Castilla-La Mancha Health Service (Other); University of Castilla-La Mancha (Other)
Responsible Party: Sponsor-Investigator, Jesús Moreno Fernández, Endocrinology and Nutrition Service, MD, PhD, Castilla-La Mancha Health Service
Organization: Castilla-La Mancha Health Service (Other)
Other Study IDs: C-127
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Results first posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-12

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Influenza Vaccines; Hepatitis B Vaccines; Vaccination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vaccination adherence: All type 1 diabetes adults patients attended in Ciudad Real General University Hospital willl be checked for Influenza Vaccination status, Pneumococcal Vaccination status and Hepatitis B Virus (HBV) status.
  Interventions: Biological: Influenza vaccination; Biological: Pneumococcal vaccination; Biological: Hepatitis B Virus (HBV) vaccination

INTERVENTIONS:
Biological: Influenza vaccination — Correct influenza vaccination status was considered in the following situation:
  - Received at least one Influenza vaccine dose in the last year.
Biological: Pneumococcal vaccination — Correct pneumococal vaccination status was considered if a subject received at least one of the following options:
  * One pneumococcal conjugate vaccine (PCV) 13 dose in the last year.
  * One PCV13 dose following a pneumococcal polysaccharide vaccine (PPSV) 23 dose between the following 8 weeks and 12 months.
  * One PPSV 23 dose in the last 5 years.
  * One PPSV23 dose in the last 5 years and a second PPSV23 dose at 5 years or PCV13 at 1 year.
Biological: Hepatitis B Virus (HBV) vaccination — Correct Hepatitis B Virus (HBV) vaccination status was considered in the following situation:
  .- Received at least three consecutive doses of HBV vaccine during six consecutive months.

SUMMARY:
Observational study about adherence to guidelines for Influenza, Pneumococcal and Hepatitis B Vaccination in adult patients with type 1 Diabetes mellitus.

DETAILED DESCRIPTION:
Cross-sectional analysis about adherence to guidelines for Influenza, Pneumococcal and Hepatitis B Vaccination in adult patients with type 1 Diabetes mellitus.

All clinical variables are gathered from two EMR softwares (Mambrino XXI and Turriano).

Data analysis is conducted using SPSS (Chicago, IL) statistics software. Results are presented as mean ± SD values or percentages. A paired Student's t-test or a Wilcoxon signed-rank test were used for the analysis of differences. Comparisons between proportions were analyzed using a chi-squared test. A P value < 0.05 was considered statistically significant.

The protocol was approved by the reference Castilla-La Mancha Public Health Institute Ethic Committee. All participants provided written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age.
* Diagnosed of Type 1 Diabetes Mellitus.
* Be attended in Ciudad Real General University Hospital.

Exclusion Criteria:

* Less than 18 years old.
* Other types of diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients attended to care in consults during this period were eligible for chart review. Patients included in the analysis were required to be ≥18 years of age and be diagnosed of type 1 diabetes mellitus.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena M Ortega Rodrigo, Study Chair — University of Castilla-La Mancha; Jose Alberto Garcia Seco, RN, Study Chair — University of Castilla-La Mancha; Fernando Garcia Seco, Study Chair — Universidad de Córdoba; Angela M Seco Segura, RN, Study Chair — Castilla-La Mancha Health Service
Locations (1):
- Obispo Rafael Torija, St., Ciudad Real, Spain

IPD SHARING:
Plan to Share IPD: Yes
In request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 year.
Access Criteria: Related investigation.

REFERENCES:
- [Background] Shah BR, Hux JE. Quantifying the risk of infectious diseases for people with diabetes. Diabetes Care. 2003 Feb;26(2):510-3. doi: 10.2337/diacare.26.2.510. PMID 12547890
- [Background] Muller LM, Gorter KJ, Hak E, Goudzwaard WL, Schellevis FG, Hoepelman AI, Rutten GE. Increased risk of common infections in patients with type 1 and type 2 diabetes mellitus. Clin Infect Dis. 2005 Aug 1;41(3):281-8. doi: 10.1086/431587. Epub 2005 Jun 16. PMID 16007521
- [Background] Alcusky MJ, Pawasauskas J. Adherence to Guidelines for Hepatitis B, Pneumococcal, and Influenza Vaccination in Patients With Diabetes. Clin Diabetes. 2015 Jul;33(3):116-22. doi: 10.2337/diaclin.33.3.116. PMID 26203204
- [Background] Sastre J, Pines PJ, Moreno J, Aguirre M, Blanco B, Calderon D, Herranz S, Roa C, Lopez J; Grupo de estudio DIACAM 1. Metabolic control and treatment patterns in patients with type 1 diabetes in Castilla-La Mancha: the DIAbetes tipo 1 in Castilla La Mancha study. Endocrinol Nutr. 2012 Nov;59(9):539-46. doi: 10.1016/j.endonu.2012.07.003. Epub 2012 Oct 4. English, Spanish. PMID 23039989
- [Background] American Association of Diabetes Educators. Vaccination practices for hepatitis B, influenza, and pneumococcal disease for people with diabetes. Diabetes Educ. 2014 Jan-Feb;40(1):122-4. doi: 10.1177/0145721713513545. No abstract available. PMID 24442103
- [Derived] Moreno-Fernandez J, Garcia-Seco JA, Rodrigo EMO, Segura AMS, Garcia-Seco F, Munoz-Rodriguez JR. Vaccination adherence to influenza, pneumococcal and hepatitis B virus in adult type 1 diabetes mellitus patients. Prim Care Diabetes. 2020 Aug;14(4):343-348. doi: 10.1016/j.pcd.2019.09.004. Epub 2019 Sep 30. PMID 31582202

RESULTS

PARTICIPANT FLOW:
Groups:
- Influenza Vaccination: All type 1 diabetes adults patients attended in Ciudad Real General University Hospital willl be checked for Influenza, Pneumococcal and HBV Vaccination status.
  Influenza vaccination: Correct influenza vaccination status was considered in the following situation:
  - Received at least one Influenza vaccine dose in the last year.
  Pneumococcal vaccination: Correct pneumococal vaccination status was considered if a subject received at least one of the following options:
  * One pneumococcal conjugate vaccine (PCV) 13 dose in the last year.
  * One PCV13 dose following a pneumococcal polysaccharide vaccine (PPSV) 23 dose between the following 8 weeks and 12 months.
  * One PPSV 23 dose in the last 5 years.
  * One PPSV23 dose in the last 5 years and a second PPSV23 dose at 5 years or PCV13 at 1 year.
  HBV vaccination: Correct HBV vaccination status was considered in the following situation:
  .- Received at least three consecutive doses of HBV vaccine during six consecutive months.
Period: Overall Study
Arm/Group | Influenza Vaccination
Started | 300
Completed | 300
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: White caucasian >18 yrs type 1 diabetes mellitus patients
Groups:
- Adherence Vaccination: All type 1 diabetes adults patients attended in Ciudad Real General University Hospital willl be checked for Influenza, pneumococcal and HBV vaccination status.
  Influenza vaccination: Correct influenza vaccination status was considered in the following situation:
  - Received at least one Influenza vaccine dose in the last year.
  Pneumococcal vaccination: Correct pneumococal vaccination status was considered if a subject received at least one of the following options:
  * One pneumococcal conjugate vaccine (PCV) 13 dose in the last year.
  * One PCV13 dose following a pneumococcal polysaccharide vaccine (PPSV) 23 dose between the following 8 weeks and 12 months.
  * One PPSV 23 dose in the last 5 years.
  * One PPSV23 dose in the last 5 years and a second PPSV23 dose at 5 years or PCV13 at 1 year.
  HBV vaccination: Correct HBV vaccination status was considered in the following situation:
  .- Received at least three consecutive doses of HBV vaccine during six consecutive months.
Arm/Group | Adherence Vaccination
Number analyzed (Participants) | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 280
  >=65 years | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160
  Male | 140
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 300
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants]
  Spain | 300

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Regional Guidelines for the Immunization of Adults With Type 1 Diabetes Mellitus (T1DM
Description: Adherence to Influenza, Pneumococcal and Hepatitis B Vaccination in adult patients with type 1 Diabetes mellitus.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Adherece Vaccination: All type 1 diabetes adults patients attended in Ciudad Real General University Hospital willl be checked for Influenza, Pneumococcal and HBV Vaccination status.
  Influenza vaccination: Correct influenza vaccination status was considered in the following situation:
  - Received at least one Influenza vaccine dose in the last year.
  Pneumococcal vaccination: Correct pneumococal vaccination status was considered if a subject received at least one of the following options:
  * One pneumococcal conjugate vaccine (PCV) 13 dose in the last year.
  * One PCV13 dose following a pneumococcal polysaccharide vaccine (PPSV) 23 dose between the following 8 weeks and 12 months.
  * One PPSV 23 dose in the last 5 years.
  * One PPSV23 dose in the last 5 years and a second PPSV23 dose at 5 years or PCV13 at 1 year.
  HBV vaccination: Correct HBV vaccination status was considered in the following situation:
  .- Received at least three consecutive doses of HBV vaccine during six consecutive months.
Arm/Group | Adherece Vaccination
Number analyzed (Participants) | 300
Participants
  influenza vaccination | 165
  Pneumoccocal vaccination | 54
  HBV vaccination | 51
  No vaccination | 30

2. Secondary Outcome: Patient Age According to Vaccination Status
Description: Age (years)
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Adherece Vaccination
Number analyzed (Participants) | 300
years
  Age : Influenzae vaccination: | 43.5 (15.2)
  Age : No influcenzae vaccination | 39.7 (13.0)
  Age : HBV vaccination | 28.3 (10.8)
  Age : HBV pneumoccocal vaccination | 44.5 (13.5)

3. Secondary Outcome: Number of Participants Who Have Taken Related Sick Leaves
Description: Number of patients who have taken related sick leaves.
Time Frame: 1 year
Measure: Number; unit: participants
Groups:
- Vaccination Adherence: All type 1 diabetes adults patients attended in Ciudad Real General University Hospital willl be checked for Influenza Vaccination status, Pneumococcal Vaccination status and Hepatitis B Virus (HBV) status.
  Influenza vaccination: Correct influenza vaccination status was considered in the following situation:
  - Received at least one Influenza vaccine dose in the last year.
  Pneumococcal vaccination: Correct pneumococal vaccination status was considered if a subject received at least one of the following options:
  * One pneumococcal conjugate vaccine (PCV) 13 dose in the last year.
  * One PCV13 dose following a pneumococcal polysaccharide vaccine (PPSV) 23 dose between the following 8 weeks and 12 months.
  * One PPSV 23 dose in the last 5 years.
  * One PPSV23 dose in the last 5 years and a second PPSV23 dose at 5 years or PCV13 at 1 year.
  Hepatitis B Virus (HBV) vaccination: Correct Hepatitis B Virus (HBV) vaccination status was considered in the following situation:
  .- Received at least three consecutive doses of HBV vaccine during six consecutive months.
Arm/Group | Vaccination Adherence
Number analyzed (Participants) | 300
participants | 17

ADVERSE EVENTS:
Time Frame: Adverse Events were not collected
Description: Adverse Events were not collected
Arm/Group | Adherence Vaccination
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-07-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT03478254/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT03478254/SAP_001.pdf
  • Informed Consent Form (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/54/NCT03478254/ICF_002.pdf